CLINICAL TRIAL: NCT03131414
Title: Inflammation, Microbiome, and Alimentation: Gastro-Intestinal and Neuropsychiatric Effects: the IMAGINE-CIHR SPOR Chronic Disease Network
Brief Title: The IMAGINE-SPOR CIHR Chronic Disease Network
Acronym: IMAGINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Paul Moayyedi, Principal Investigator, Hamilton Health Sciences Corporation
Other Study IDs: REB#3000
Record Dates: First submitted 2017-03-10; First posted 2017-04-27 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: IBS - Irritable Bowel Syndrome; Ulcerative Colitis; Crohn Disease; Healthy
MeSH Terms: conditions — Irritable Bowel Syndrome; Colitis, Ulcerative; Crohn Disease | interventions — Diet; Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Irritable bowel syndrome: A total of 2000 patients with IBS who have met Rome IV criteria are 13 years of age or older will be consented and recruited for this study.
  IBS patients will be categorized into diarrhea predominant IBS (IBS-D), constipation predominant IBS (IBS-C) or alternating constipation and diarrhea (IBS-A) or unclassified IBS (IBS-U). A detailed diet history will be obtained and gastrointestinal microbiome will be evaluated.
  Interventions: Other: Diet; Other: Gastrointestinal microbiome
- Ulcerative colitis: 2000 CD and 2000 UC cases over the age of 4 years will be enrolled.
  Montreal Classification will be used for adult UC patients, and the Paris classification for pediatric UC. The research coordinator will conduct a chart review to confirm date of diagnosis and maximal phenotype at time of enrolment. A detailed diet history will be obtained and gastrointestinal microbiome will be evaluated.
  Interventions: Other: Diet; Other: Gastrointestinal microbiome
- Crohn's disease: 2000 CD cases over the age of 4 years will be enrolled.
  Montreal Classification will be used for adult CD patients, and the Paris classification for pediatric CD. The research coordinator will conduct a chart review to confirm date of diagnosis and maximal phenotype at time of enrolment. A detailed diet history will be obtained and gastrointestinal microbiome will be evaluated.
  Interventions: Other: Diet; Other: Gastrointestinal microbiome
- Healthy control: A total of 2000 healthy family members, relative or friends of cohort participants over the age of 4 will be consented and recruited for this study.
  Each control that agrees to participate will undergo an initial screening questionnaire to confirm that they are healthy and have no gastrointestinal symptoms using the ROME IV Questionnaire. A detailed diet history will be obtained and gastrointestinal microbiome will be evaluated.
  Interventions: Other: Diet; Other: Gastrointestinal microbiome

INTERVENTIONS:
Other: Diet — Dietary intake
Other: Gastrointestinal microbiome — Genomic sequencing of stool for gut bacteria

SUMMARY:
The IMAGINE Cohort Study will identify and recruit a cohort of 8000 patients with IBS, IBD and healthy controls (2000 of each) who will be assessed in terms of their psychological status, dietary intake, gut microbiome, metabolomic and inflammatory markers and genotype, health-related quality of life, and health care resource use and associated costs. The cohort and healthy controls will be followed prospectively for up to 5 years after the completion of study enrolment.

DETAILED DESCRIPTION:
The goal of the screening visit is to confirm that the Subject/Healthy Control is willing to participate in the study and that they meet the eligibility criteria for the study.

The screening visit will include:

i. Obtaining signed informed consent /assent to screen for eligibility (Consent/Assent-Subject, Consent/Assent-Control).

ii. Reviewing the subject/control for eligibility (per inclusion/exclusion criteria).

Subjects will be identified through several pathways: 1) Patients with confirmed IBS or IBD in existing site databases who have previously consented to be contacted for future IBS studies or those approached in clinic with a recent confirmed diagnosis of IBS/IBD and consent to participate and 2) patients with self-reported IBS or IBD who contact the site coordinator or who are identified in clinic with an unsubstantiated diagnosis of IBS/IBD.

Subjects with a confirmed diagnosis of IBS or IBD and who have given prior consent to be contacted, will be prescreened by phone or in person. All others will be invited to a screening visit and the study rationale and design will be explained. Interested subjects will be asked to provide informed written consent. Eligibility will then be confirmed and subjects will complete the questionnaires and provide the necessary samples at this and a follow-up visit if necessary.

Subjects who do not meet the diagnostic criteria for IBS or IBD and wish to have the diagnosis confirmed, will be advised to see their family physician for any necessary diagnostic testing. A letter to the family physician will be provided stating that the patient had been approached about the study and that the diagnosis of IBS/IBD could not been made due to an absence of testing and/or failure to meet the predefined criteria. Patients will also be informed if they fail to meet other eligibility criteria that would exclude them from the study.

When eligibility for subjects and healthy controls has been confirmed, the following questionnaires will be answered and samples obtained:

* Blood samples
* Metabolomic urine sample
* Stool sample (metagenomics, metabolomics, fecal calprotectin (FCAL) and β-defensins)
* Demographic questionnaire
* Quality of life questionnaire (EQ-5D for adults)
* Food Frequency Questionnaire
* Psychological questionnaires (pediatric for ≤ 17 years, adult for those > 17 years)
* Optional on-line additional psychological questionnaires for adults
* Disease specific questionnaires (UC, CD and IBS - UC and CD further divided into pediatric for ≤ 17 years, adult for those > 17 years)
* General gastrointestinal symptom questionnaires (Short for Leeds Dyspepsia Questionnaire, PROMIS diarrhea, PROMIS abdominal pain, PROMIS constipation and PROMIS bloating).
* Workplace productivity questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Each control that agrees to participate will undergo an initial screening questionnaire to confirm that they are healthy and have no gastrointestinal symptoms using the ROME IV Questionnaire.

Exclusion Criteria:

* • major gastrointestinal surgery (Roux en y, bowel resection)

  * any major comorbid chronic condition (e.g. decompensated liver disease or malignancy, lung or cardiac disease, active HIV, diabetes mellitus requiring medication,
  * difficulties with communication or conditions affecting ability to provide informed consent,
  * unable to communicate in the language of the cohort study (English or French)
  * those who do not wish to participate in this study
  * diagnosis of schizophrenia
  * diagnosis of eating disorder

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There will be 17 recruitment centres across Canada responsible for recruitment of 2000 subjects with CD, 2000 subjects with UC, 2000 subjects with IBS and 2000 healthy controls. Each centre will be required to obtain appropriate ethics approval prior to initiating study recruitment.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
IMAGINE microbiome and diet | baseline
  Microbiome and dietary comparison between UC, CD, IBS and controls predictors of failure of therapy (each class of therapy in UC, CD, IBS and each disease will be analyzed separately)

SECONDARY OUTCOMES:
IMAGINE metabolomics | baseline and five years
  Metabolomic comparison between UC, CD, IBS and controls
IMAGINE anxiety | baseline and five years
  Anxiety score evaluated using PROMIS questionnaire between UC, CD, IBS and controls
IMAGINE depression | baseline and five years
  Depression score evaluated using PROMIS questionnaire between UC, CD, IBS and controls
IMAGINE health related costs | baseline and five years
  Health related costs measured by provincial databases and questionnaire between UC, CD, IBS and controls
IMAGINE microbiome and diet | five years
  Microbiome and dietary comparison between UC, CD, IBS and controls

CONTACTS AND LOCATIONS:
Overall Officials: Paul Moayyedi, MD, Principal Investigator — HHSC
Locations (1):
- Hamilton Health Sciences / McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moayyedi P, MacQueen G, Bernstein CN, Vanner S, Bercik P, Madsen KL, Surette M, Rioux JD, Dieleman LA, Verdu E, de Souza RJ, Otley A, Targownik L, Lavis J, Cunningham J, Marshall DA, Zelinsky S, Fernandes A. IMAGINE Network's Mind And Gut Interactions Cohort (MAGIC) Study: a protocol for a prospective observational multicentre cohort study in inflammatory bowel disease and irritable bowel syndrome. BMJ Open. 2020 Oct 21;10(10):e041733. doi: 10.1136/bmjopen-2020-041733. PMID 33087380